CLINICAL TRIAL: NCT07401680
Title: A Multi-centre, Randomised Controlled Trial Comparing Fecal Microbiota Transplantation to Placebo in an Expanded Ulcerative Colitis Population: a Feasibility Study (FRONTIER-UC)
Brief Title: Fecal Microbiota Transplantation in an Expanded Ulcerative Colitis Population
Acronym: FRONTIER-UC
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pro00160199
Record Dates: First submitted 2026-01-27; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ulcerative Colitis; Inflammatory Bowel Diseases; Clostridioides Difficile Infection
Keywords: Fecal microbiota transplantation; FMT; Lyophilized fecal microbiota transplantation; LFMT
MeSH Terms: conditions — Colitis, Ulcerative; Inflammatory Bowel Diseases; Clostridium Infections

STUDY DESIGN:
Intervention Model Description: Multi-center, randomized, double-blind, placebo-controlled feasibility study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Adjunct therapy group (LFMT) (Experimental): Induction phase: 4 capsules a day x 1 week, 2 capsules a day x 1 week, followed by 1 capsule daily x 6 weeks
  Maintenance phase: 1 capsule daily x 16 weeks
  Interventions: Other: Lyophilized Fecal Microbiota Transplantation (LFMT)
- Adjunct therapy group (Placebo) (Placebo Comparator): The placebo capsules will appear identical to LFMT capsules and same dosing will apply.
  Interventions: Other: Placebo
- Co-Administration therapy group (LFMT) (Experimental): Induction phase: 4 capsules a day x 1 week, 2 capsules a day x 1 week, followed by 1 capsule daily x 6 weeks
  Maintenance phase: 1 capsule daily x 16 weeks
  Interventions: Other: Lyophilized Fecal Microbiota Transplantation (LFMT)
- Co-Administration therapy group (Plcebo) (Placebo Comparator): The placebo capsules will appear identical to LFMT capsules and same dosing will apply.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Lyophilized Fecal Microbiota Transplantation (LFMT) — LFMT by oral capsules
  Arms: Adjunct therapy group (LFMT); Co-Administration therapy group (LFMT)
Other: Placebo — Placebo capsules does not contain FMT
  Arms: Adjunct therapy group (Placebo); Co-Administration therapy group (Plcebo)

SUMMARY:
This is a multi-centre, randomised controlled trial comparing fecal microbiota transplantation to placebo in an expanded ulcerative colitis population: a feasibility study (FRONTIER-UC) to determine whether a full-scale randomized controlled trial (RCT) to investigate fecal microbiota transplantation (FMT) in ulcerative colitis (UC) is feasible.

DETAILED DESCRIPTION:
This is a randomized, double blind, placebo-controlled trial for UC patients with active disease.

Participants will be grouped into one of two categories

1. Add to current therapy (i.e., adjunct therapy)

   or
2. Initiate or switch to a new advanced agent (i.e., co-administration)

The study will recruit 85 outpatients at 3 Canadian healthcare centres

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Able to provide informed consent
3. Established UC diagnosis through standard endoscopic and histologic criteria
4. Active UC
5. Use of effective contraception method for women of childbearing potential for at least 4 weeks prior to receiving study treatment and for the duration of the trial
6. Willing and able to comply with all required study procedures

Exclusion Criteria:

1. Severe UC requiring hospitalization
2. Crohn's disease or indeterminate colitis
3. Irritable bowel syndrome
4. Intestinal infection within 4 weeks of enrollment
5. Evidence of toxic megacolon or gastrointestinal perforation on imaging
6. Planned colectomy
7. Abdominal surgery within 60 days of enrollment
8. Neutropenia with absolute neutrophil count <0.5 x 109/L
9. Peripheral white blood cell count > 35.0 x 109/L and fever (>38C)
10. Planned or actively taking another investigational product
11. Uncontrolled medical conditions such as psychiatric disorders or substance abuse
12. Severe underlying disease such that the patient is not expected to survive for at least 30 days
13. Pregnancy or breastfeeding
14. Unwilling to discontinue non-dietary probiotic
15. Antibiotic use 30 days prior to enrollment or anticipated need for systemic antibiotic use during study
16. FMT for any reason within 6 months of enrollment
17. Investigator's judgement that enrolment is not in the best interest of the patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-12-01 (Estimated)

PRIMARY OUTCOMES:
Steroid-free endoscopic remission | At 8 weeks
  Steroid-free endoscopic remission is defined as either
  1. Mayo endoscopy score (MES)= 0 OR
  2. MES=1 + FC <150 µg/g

SECONDARY OUTCOMES:
Serious adverse events [SAE] | up to week 24 or at time of withdrawal
  SAEs including infections attributable to FMT, hospitalization due to UC exacerbation or complications related to FMT, or colectomy due to UC
Adverse outcomes | up to week 24 or upon withdrawal
  Adverse outcomes, including nausea, vomiting, worsening diarrhea or abdominal pain
Quality of Life- sIBDQ | Baseline to 8 weeks and 24 weeks
  Changes in health-related quality of life measures using the short IBD questionnaire (sIBDQ)
Quality of Life- WPAI-IBD | Baseline to 8 weeks and weeks 24
  Changes in health-related quality of life measures using the work productivity and activity impairment questionnaire (WPAI-IBD)

OTHER OUTCOMES:
Recruitment rate | Study start to the end of recruitment
  Evaluation of rate of participant recruitment
Consent rate | Study start to the end of recruitment
  Evaluation of rate of participant consent to participate
Symptom remission | 8 weeks and 24 weeks
  Symptom remission, defined as partial Mayo score <2 with no individual subscore >1
Symptom response | At weeks 8 and 24
  Symptom response, defined as reduction in partial Mayo score by >2 points from baseline and >30% from baseline and decrease in rectal bleeding score >1 point from baseline
Endoscopic improvement | At week 8 and 24
  Endoscopic improvement, defined as a decrease of Mayo endoscopy score (MES) by at least 1 point
UC therapy escalation | At weeks 8 and 24
  Avoidance of UC therapy escalation
Stool microbial compositions | between week 0 to 8 weeks and week 0 to 24 weeks
  Changes in stool microbial compositions

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta

IPD SHARING:
Plan to Share IPD: No